CLINICAL TRIAL: NCT04555733
Title: An Open-Label, Single and Multiple Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Lemborexant in Healthy Chinese Subjects
Brief Title: A Single and Multiple Dose Study of Lemborexant in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E2006-J086-014
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2020-09

CONDITIONS: Healthy Volunteer
Keywords: Pharmacokinetics; Phase 1; E2006; Healthy Participants
MeSH Terms: interventions — lemborexant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Lemborexant 5 mg (Experimental): Participants will receive a single dose of lemborexant 5 milligram (mg) tablet, orally on Day 1.
  Interventions: Drug: Lemborexant
- Cohort 2: Lemborexant 10 mg (Experimental): Participants will receive a single dose of lemborexant 10 mg tablet, orally on Day 1 followed by a washout period of approximately 14 days further followed by multiple doses of lemborexant 10 mg tablets, orally, once daily from Day 15 through Day 28.
  Interventions: Drug: Lemborexant
- Cohort 3: Lemborexant 25 mg (Experimental): Participants will receive a single dose of lemborexant 25 mg (1*5 mg tablet and 2*10 mg tablet), orally on Day 1.
  Interventions: Drug: Lemborexant

INTERVENTIONS:
Drug: Lemborexant — Lemborexant oral tablets.
  Other Names: E2006; Dayvigo

SUMMARY:
The primary objective of this study is to assess the pharmacokinetics (PK) of lemborexant and metabolites (M4, M9, and M10) in plasma in healthy Chinese participants following single and multiple oral doses of lemborexant.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese adult male or female participants living in China.
2. Non-smoking, age greater than or equal to (>=) 18 years and less than or equal to (<=) 45 years old at the time of obtaining written consent. To be considered non-smokers, participant must have discontinued smoking for at least 4 weeks before first dosing.
3. Participants with a body mass index (BMI) of 19 to 24 kilogram per square meter (kg/m^2) at screening.

Exclusion Criteria:

1. Participants who weigh less than 50 kilogram (kg) at Screening.
2. Females who are breastfeeding or pregnant (as documented by a positive beta-human chorionic gonadotropin [β-hCG] test with a minimum sensitivity of International units per liter (IU/L) or equivalent units of β-hCG). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
3. Females of childbearing potential who:

   a. Within 28 days before study entry, did not use a highly effective method of contraception, which includes any of the following:

   i. total abstinence (if it is their preferred and usual lifestyle)

   ii. an intrauterine device or intrauterine hormone-releasing system (IUS)

   iii. a contraceptive implant

   iv. an oral contraceptive except for contraceptives containing levonorgestrel (with additional barrier method) (Participant must be on a stable dose of the same oral contraceptive product for at least 28 days before dosing and throughout the study and for 28 days after study drug discontinuation.)

   v. have a vasectomized partner with confirmed azoospermia.

   b. Do not agree to use a highly effective method of contraception (as described above) throughout the entire study period and for 28 days after study drug discontinuation.

   It is permissible that if a highly effective method of contraception is not appropriate or acceptable to the participant, then the participant must agree to use a medically acceptable method of contraception, that is, double-barrier methods of contraception such as latex or synthetic condom plus diaphragm or cervical/vault cap with spermicide.

   NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (that is, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
4. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks before first dosing.
5. Evidence of disease that may influence the outcome of the study within 4 weeks before first dosing; example psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism.
6. Any suicidal ideation with intent to act with or without a plan at screening or within 6 months of screening.
7. Any suicidal behavior within 10 years of screening.
8. Any history of gastrointestinal surgery that may affect PK profiles of lemborexant, example, hepatectomy, digestive organ resection at screening.
9. Any clinically abnormal symptom or organ impairment based on medical history, physical examination, vital signs, electrocardiogram (ECG) or laboratory test results, which require medical treatment.
10. A prolonged QT/QTc interval (QT interval corrected for heart rate by Fridericia's formula [QTcF] greater than (>) 450 milliseconds [ms]) as demonstrated by a repeated ECG.
11. Known history of clinically significant drug allergy at Screening.
12. Known history of food allergy or presently experiencing significant seasonal or perennial allergy at Screening.
13. Human immunodeficiency virus (HIV) positive demonstrated by positive serology at Screening.
14. Active viral hepatitis (B or C) as demonstrated by positive serology at Screening.
15. History of drug or alcohol dependency or abuse within 2 years before Screening, or a positive urine drug test or breathe alcohol test.
16. Participants who contravene the restrictions on concomitant medications, food and beverages during the Screening Period.
17. Currently enrolled in another clinical study or used any investigational drug or device within 28 days or 5 half-lives, whichever is longer, preceding informed consent.
18. Receipt of blood products within 4 weeks, or donation of blood or plasma within 3 months before first dosing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for Lemborexant and Its Metabolites (M4, M9, and M10) Following Single Dose in All Cohorts | All Cohorts, Day 1: 0-240 hours post single dose
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Lemborexant and Its Metabolites (M4, M9, and M10) Following Single Dose in All Cohorts | All Cohorts, Day 1: 0-240 hours post single dose
AUC(0-8h): Area Under the Concentration-time Curve From Zero Time to 8 Hours Postdose for Lemborexant and Its Metabolites (M4, M9, and M10) Following Single Dose in All Cohorts | All Cohorts, Day 1: 0-8 hours post single dose
AUC(0-24h): Area Under the Concentration-time Curve From Zero Time to 24 Hours Postdose for Lemborexant and Its Metabolites (M4, M9, and M10) Following Single Dose in All Cohorts | All Cohorts, Day 1: 0-24 hours post single dose
AUC(0-t): Area Under the Concentration-time Curve From Zero Time to Time of Last Quantifiable Concentration for Lemborexant and Its Metabolites (M4, M9, and M10) Following Single Dose in All Cohorts | All Cohorts, Day 1: 0-240 hours post single dose
AUC(0-inf): Area Under the Concentration-time Curve From Zero Time Extrapolated to Infinite Time for Lemborexant and Its Metabolites (M4, M9, and M10) Following Single Dose in All Cohorts | All Cohorts, Day 1: 0-240 hours post single dose
λz: Terminal Phase Rate Constant for Lemborexant and Its Metabolites (M4, M9, and M10) Following Single Dose in All Cohorts | All Cohorts, Day 1: 0-240 hours post single dose
t½: Terminal Elimination Phase Half-life for Lemborexant and Its Metabolites (M4, M9, and M10) Following Single Dose in All Cohorts | All Cohorts, Day 1: 0-240 hours post single dose
MRT: Mean Residence Time for Lemborexant and Its Metabolites (M4, M9, and M10) Following Single Dose in All Cohorts | All Cohorts, Day 1: 0-240 hours post single dose
Vz/F: Apparent Volume of Distribution at Terminal Phase for Lemborexant Following Single Dose in All Cohorts | All Cohorts, Day 1: 0-240 hours post single dose
CL/F: Apparent Total Clearance Following Extravascular Administration for Lemborexant Following Single Dose in All Cohorts | All Cohorts, Day 1: 0-240 hours post single dose
Metabolite to Lemborexant Area Under the Concentration-time Curve From Zero Time Extrapolated to Infinite Time Ratio Following Molecular Weight Correction to Lemborexant Equivalents After Single Dose in All Cohorts | All Cohorts, Day 1: 0-240 hours post single dose
Cmax: Maximum Observed Plasma Concentration for Lemborexant and Its Metabolites (M4, M9, and M10) Following Single Dose (Day 15 dosing) in Cohort 2 | Cohort 2, Day 15: 0-24 hours post single dose
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Lemborexant and Its Metabolites (M4, M9, and M10) Following Single Dose (Day 15 dosing) in Cohort 2 | Cohort 2, Day 15: 0-24 hours post single dose
AUC(0-8h): Area Under the Concentration-time Curve From Zero Time to 8 Hours Postdose for Lemborexant and Its Metabolites (M4, M9, and M10) Following Single Dose (Day 15 dosing) in Cohort 2 | Cohort 2, Day 15: 0-8 hours post single dose
AUC(0-24h): Area Under the Concentration-time Curve From Zero Time to 24 Hours Postdose for Lemborexant and Its Metabolites (M4, M9, and M10) Following Single Dose (Day 15 dosing) in Cohort 2 | Cohort 2, Day 15: 0-24 hours post single dose
AUC(0-8h): Area Under the Concentration-time Curve From Zero Time to 8 Hours Postdose for Lemborexant and Its Metabolites (M4, M9, and M10) Following Multiple Doses (Day 28 dosing) in Cohort 2 | Cohort 2, Day 28: 0-8 hours post multiple dose
AUC(0-τ): Area Under the Concentration-time Curve Over the Dosing Interval for Lemborexant and Its Metabolites (M4, M9, and M10) Following Multiple Doses in Cohort 2 | Cohort 2, Day 28: 0-324 hours post multiple dose
Css,avg: Average Steady State Concentration for Lemborexant and Its Metabolites (M4, M9, and M10) Following Multiple Doses in Cohort 2 | Cohort 2, Day 28: 0-324 hours post multiple dose
Css,max: Maximum Observed Concentration at Steady State for Lemborexant and Its Metabolites (M4, M9, and M10) Following Multiple Doses in Cohort 2 | Cohort 2, Day 28: 0-324 hours post multiple dose
Css,min: Minimum Observed Concentration at Steady State for Lemborexant and Its Metabolites (M4, M9, and M10) Following Multiple Doses in Cohort 2 | Cohort 2, Day 28: 0-324 hours post multiple dose
PTF: Peak-trough Fluctuation for Lemborexant and Its Metabolites (M4, M9, and M10) Following Multiple Doses in Cohort 2 | Cohort 2, Day 28: 0-324 hours post multiple dose
Tss,max: Time to Reach the Maximum Plasma Concentration (Cmax) for Lemborexant and Its Metabolites (M4, M9, and M10) Following Multiple Doses at Steady State in Cohort 2 | Cohort 2, Day 28: 0-324 hours post multiple dose
λz: Terminal Phase Rate Constant for Lemborexant and Its Metabolites (M4, M9, and M10) Following Multiple Doses in Cohort 2 | Cohort 2, Day 28: 0-324 hours post multiple dose
t½: Terminal Elimination Phase Half-life for Lemborexant and Its Metabolites (M4, M9, and M10) Following Multiple Doses in Cohort 2 | Cohort 2, Day 28: 0-324 hours post multiple dose
MRT: Mean Residence Time for Lemborexant and Its Metabolites (M4, M9, and M10) Following Multiple Doses in Cohort 2 | Cohort 2, Day 28: 0-324 hours post multiple dose
Vz/F: Apparent Volume of Distribution at Terminal Phase for Lemborexant Following Multiple Doses in Cohort 2 | Cohort 2, Day 28: 0-324 hours post multiple dose
CLss/F: Apparent Total Clearance Following Extravascular Administration at Steady-state for Lemborexant Following Multiple Doses in Cohort 2 | Cohort 2, Day 28: 0-324 hours post multiple dose
Rac: Accumulation Ratio for Lemborexant and Its Metabolites (M4, M9, and M10) Following Multiple Doses in Cohort 2 | Cohort 2, Day 28: 0-324 hours post multiple dose
Metabolite to Lemborexant Area Under the Concentration-time Curve Over the Dosing Interval Ratio Following Molecular Weight Correction to Lemborexant Equivalents After Multiple Doses in Cohort 2 | Cohort 2, Day 28: 0-324 hours post multiple dose

CONTACTS AND LOCATIONS:
Locations (1):
- Xuhui Central Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.